CLINICAL TRIAL: NCT01971294
Title: Lower Urinary Tract Symptoms in Patients Suffering From Systemic Sclerosis: a Multi-centric Longitudinal Study
Brief Title: Lower Urinary Tract Symptoms in Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University Hospital, Paris (Other); Azienda Ospedaliera di Padova (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Gregor John, Gregor John, University Hospital, Geneva
Other Study IDs: CER 12-291
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Urinary Symptoms; Systemic Sclerosis
Keywords: Urinary symptoms; Systemic sclerosis; Severity index; Urinary tract infection; mortality; Quality of life
MeSH Terms: conditions — Scleroderma, Systemic; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Systemic sclerosis: Adult suffering from systemic sclerosis included in the EUSTAR network of Brescia (I), Geneva (CH), Padova (I) and Paris (F).

SUMMARY:
Urinary symptoms must be frequent in Scleroderma. In one hand, mobility limitation by joint stiffness and skin sclerosis, forced diuresis due to heart involvement (cardiomyopathy or pulmonary hypertension), diuretics use and corticoid-induced hyperglycaemia, as well as narcotic medication use, puts patients at higher risk of secondary bladder filling and voiding dysfunction. In another hand, few case report and small sample observational studies have identified a specific sclerosis of the urinary tract. Those two mechanisms must be more frequent in the diffuse cutaneous form of scleroderma (dcSSc) compare to the limited one (lcSSc). But prevalence or incidence is unknown.

Urinary symptoms are seldom reported by those suffering from them and are rarely part of a systemic evaluation. In a threatening disease, urinary symptoms assessment might seem to be of no priority. But LUTS have a real impact on many aspect of everyday living. Furthermore urinary tract involvement might predispose to urinary tract infection due to flow limitation and stagnation. Since it is an inner fibrosis it might be associated with a more aggressive form of disease conferring a greater loss of physical function, higher risk for hospital admission and death.

Thus, identifying urinary symptoms would permit to address specific rehabilitation or medication therapy, in order to minimize the consequences of the bothersome symptoms and identify those subjects at higher risk of urinary infection, aggressive disease/loss of function or death.

This study will also give basement to build an interventional study directed toward LUTS treatment in this population.

In this prospective cohort we would like to:

* Compare the prevalence of lower urinary tract symptoms (LUTS) in diffuse and limited forms of systemic sclerosis.
* Determine the prevalence (at inclusion) and incidence (in a two years period) of LUTS among patients suffering from systemic sclerosis.
* Evaluate the impact of LUTS symptoms on Quality of life.
* Compare the discrimination ability of Cochin-hand score and HAQ score to predict incontinence in this population.
* Evaluate the association between LUTS symptoms, hospital admission rate, urinary tract infection, mortality and loss of autonomy.

ELIGIBILITY:
Inclusion Criteria:

Adult suffering from systemic sclerosis included in network of Brescia (I), Geneva (CH), Padova (I) and Paris (F).

Exclusion Criteria:

Those unable to understand the rules and implications of the study, end of life patients, the pregnant women and anuric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systemic sclerosis suffering patients in Brescia (I), Geneva (CH), Padova (I) and Paris (F)
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Prevalence/incidence of urinary symptoms in scleroderma | Inclusion and every year for 2 years

SECONDARY OUTCOMES:
Short Form 36 Health Survey (SF-36) | At inclusion and after 2 years
  Quality of life (lower, better)
Mortality | During two years
Urinary tract infection | During two years
Incontinence Quality of Life (IQol) | At inclusion and after 2 years
  Quality of life (0-100; higher, better), specific for urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Chizzolini, Pr, Study Director — University Hospital, Geneva; Yannick Allanor, Pr, Study Chair — Département de médecine interne, Hôpital Cochin, Paris; Franco Cozzi, MD, Study Chair — Department of Rheumatology, Azienda Ospedaliera di Padova, Padova (I); Paolo Airo, MD, Study Chair — Department of Rheumatology and Clinical Immunology, Azienda Ospedaliera Spedali Civili di Brescia, Brescia (I); Franco Franceschini, MD, Study Chair — Department of Rheumatology and Clinical Immunology, Azienda Ospedaliera Spedali Civili di Brescia, Brescia (I)
Locations (4):
- Hôpital Cochin, Paris, France
- Italy (2):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera di Padova, Padua
- Universtiy Hospital, Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] John G, Avouac J, Piantoni S, Polito P, Fredi M, Cozzi F, Airo P, Truchetet ME, Franceschini F, Allanore Y, Chizzolini C. Prevalence and Disease-Specific Risk Factors for Lower Urinary Tract Symptoms in Systemic Sclerosis: An International Multicenter Study. Arthritis Care Res (Hoboken). 2018 Aug;70(8):1218-1227. doi: 10.1002/acr.23454. Epub 2018 Jun 19. PMID 29073343
- [Derived] John G, Allanore Y, Polito P, Piantoni S, Fredi M, Avouac J, Franceschini F, Truchetet ME, Cozzi F, Airo P, Chizzolini C. The limited cutaneous form of systemic sclerosis is associated with urinary incontinence: an international multicentre study. Rheumatology (Oxford). 2017 Nov 1;56(11):1874-1883. doi: 10.1093/rheumatology/kex230. PMID 28977630